CLINICAL TRIAL: NCT03680755
Title: Efficacy of an Internet-based Intervention for Dental Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U01DE027328 (NIH); U01DE027328 (NIH)
Record Dates: First submitted 2018-08-30; First posted 2018-09-21 (Actual); Results first posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Dental Anxiety
Keywords: dental avoidance; dental phobia; pain sensitivity

STUDY DESIGN:
Intervention Model Description: This will be a single-center parallel groups study with randomization to one of three arms: (1) a treatment condition (Tr1) in which the dental anxiety intervention is administered by CBT personnel (n=150), (2) a treatment condition in which the dental anxiety intervention is administered by dental staff (Tr2) (n=150), or (3) an active control (AC) group (notification of the dental providers of the patient's score on a dental anxiety scale before their dental treatment appointment). In addition, control participants will be asked to view a video of nature scenes for a period of time equivalent to the dental anxiety intervention.
Masking Description: Given the obvious differences between those who will receive the Internet-based dental anxiety and those who will not (i.e., those who are assigned to the control condition), we will not be able to blind patients to this aspect of randomization. Patients will not be informed about the professional affiliation of therapy aides, who will dress similarly (e.g., professional dress and a lab coat) and who will be instructed not to respond to questions related to this topic.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tr1 group (Experimental): Participants assigned to Tr1 will complete the experimental dental anxiety management program, which will be facilitated by a person trained in psychological treatments. This program consists of a series of videos which provide information about dental anxiety, educate about the details of three dental procedures which are anxiety-provoking for the participant, and teach them how to cope better with the dental experience. This program will take about 60 minutes to complete.
  Interventions: Behavioral: Internet-based intervention for dental anxiety
- Tr2 group (Experimental): Participants assigned to Tr2 will complete the experimental dental anxiety management program, which will be facilitated by dental staff. This program consists of a series of videos which provide information about dental anxiety, educate about the details of three dental procedures which are anxiety-provoking for the participant, and teach them how to cope better with the dental experience. This program will take about 60 minutes to complete.
  Interventions: Behavioral: Internet-based intervention for dental anxiety
- Active control (No Intervention): Participants assigned to the control group, will not complete the experimental dental anxiety management program at this time. They will complete study paperwork and watch a non-dental video for 45 minutes before their scheduled dental appointment. Immediately after the dental appointment, they will complete a brief interview with the research staff person.

INTERVENTIONS:
Behavioral: Internet-based intervention for dental anxiety — Participants will complete the experimental dental anxiety management program, which will be facilitated by a person trained in psychological treatments or by dental staff. This program consists of a series of videos which provide information about dental anxiety, educate about the details of three dental procedures which are anxiety-provoking for the participant, and teach them how to cope better with the dental experience. This program will take about 60 minutes to complete.
  Arms: Tr1 group; Tr2 group

SUMMARY:
The overall objective of the activities described in this protocol is to examine the efficacy of the Internet-based intervention in the reduction of dental anxiety in patients seeking dental treatment. This study has 2 primary objectives and 2 secondary objectives:

Primary Objective 1-Therapy Aides: To compare the efficacy of the intervention as administered by personnel with training and experience in cognitive behavioral therapy (CBT) to the efficacy of the intervention as administered by dental staff who have undergone a brief but specific training in the administration of the intervention.

Primary Objective 2-Intervention Efficacy: To compare the efficacy of the intervention, administered by either type of therapy aide (CBT personnel or dental staff), to an active control condition.

Secondary Objective 1-Tests of Moderators: To examine whether baseline levels of distress tolerance and pain sensitivity moderate the efficacy of the dental anxiety intervention, regardless of therapy aide, in comparison to an active control condition.

Secondary Objective 2-Other Intervention Effects: To explore effects of the intervention beyond primary efficacy, including attendance at recall visits in the 12 months after the intervention; pain intensity; avoidance due to fear of dental procedures; and client satisfaction.

DETAILED DESCRIPTION:
This clinical trial will evaluate the efficacy of a brief Internet-based cognitive-behavioral intervention for the treatment of impairing dental anxiety among those seeking dental care at the clinics of a university dental school. The primary objective of human subjects activities described in this protocol is to evaluate the efficacy of the Internet-based intervention for dental anxiety among patients presenting to the participating clinic(s). To achieve this overall objective, 2 primary objectives and 2 secondary objectives have been proposed:

Primary Objective 1-Therapy Aides: To compare the efficacy of the intervention as administered by personnel with training and experience in cognitive behavioral therapy (CBT) to the efficacy of the intervention as administered by dental staff who have undergone a brief but specific training in the administration of the intervention. Efficacy will be indexed by measures of dental anxiety and fear completed at 1-month and 3-month follow-up assessments.

Primary Objective 2-Intervention Efficacy: To compare the efficacy of the intervention, administered by either type of therapy aide (CBT personnel or dental staff), to an active control condition. Efficacy will be indexed by measures of dental anxiety and fear completed at 1-month and 3-month follow-up assessments.

Secondary Objective 1-Tests of Moderators: To examine whether baseline levels of distress tolerance and pain sensitivity moderate the efficacy of the dental anxiety intervention, regardless of therapy aide, in comparison to an active control condition.

Secondary Objective 2-Other Intervention Effects: To explore effects of the intervention beyond primary efficacy, including attendance at recall visits in the 12 months after the intervention; pain intensity; avoidance due to fear of dental procedures; and client satisfaction.

Patients (N=450) between the ages of 18 and 75 attending the Temple University Kornberg School of Dentistry (TUKSoD) dental clinics and reporting high dental anxiety that causes at least mild impairment will be recruited and consented. To obtain the sample, the investigators will screen all patients who present to the Faculty Practice Clinic (FPC) of TUKSoD (as well as the Graduate Clinics of TUKSoD [Endodontology, Periodontology, Advanced Education General Dentistry], if necessary). Total participation time for each patient is approximately 4 months but could be slightly longer pending the interval between screening/baseline and the scheduled date of the dental anxiety intervention/dental appointment.

ELIGIBILITY:
Inclusion Criteria:

* patient endorses high dental anxiety (a score of 19 or a score of 4-5 on at least 2 of the 5 items) on the MDAS
* endorses at least mild impairment as a result of that anxiety at the baseline interview as indexed by the appropriate rating in the specific phobia module of the ADIS-5
* be between 18 and 75 years of age
* be sufficiently fluent in written and spoken English in the judgment of project staff that the patient would be able to benefit from the intervention and validly complete the assessments.

Exclusion Criteria:

* a self-reported current medical condition (e.g., cardiopulmonary disease, seizure disorder) that might make exposure to anxiety-evoking stimuli inadvisable
* current suicidal/homicidal ideation/intent or other condition that would take priority over an intervention focused on dental anxiety
* current psychosis, mental retardation, or other condition that would significantly diminish the patient's ability to adequately focus attention adaptively on the current protocol
* inability to give informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2024-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marisol Tellez Merchan, PhD, Principal Investigator — Professor; Eugene M Dunne, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Maurice H Kornberg School of Dentistry Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Humphris GM, Morrison T, Lindsay SJ. The Modified Dental Anxiety Scale: validation and United Kingdom norms. Community Dent Health. 1995 Sep;12(3):143-50. PMID 7584581
- [Background] Brahm CO, Lundgren J, Carlsson SG, Nilsson P, Corbeil J, Hagglin C. Dentists' views on fearful patients. Problems and promises. Swed Dent J. 2012;36(2):79-89. PMID 22876395
- [Background] Farrar JT, Polomano RC, Berlin JA, Strom BL. A comparison of change in the 0-10 numeric rating scale to a pain relief scale and global medication performance scale in a short-term clinical trial of breakthrough pain intensity. Anesthesiology. 2010 Jun;112(6):1464-72. doi: 10.1097/ALN.0b013e3181de0e6d. PMID 20463579
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Gordon D, Heimberg RG, Tellez M, Ismail AI. A critical review of approaches to the treatment of dental anxiety in adults. J Anxiety Disord. 2013 May;27(4):365-78. doi: 10.1016/j.janxdis.2013.04.002. Epub 2013 Apr 13. PMID 23746494
- [Background] Tellez M, Potter CM, Kinner DG, Jensen D, Waldron E, Heimberg RG, Myers Virtue S, Zhao H, Ismail AI. Computerized Tool to Manage Dental Anxiety: A Randomized Clinical Trial. J Dent Res. 2015 Sep;94(9 Suppl):174S-80S. doi: 10.1177/0022034515598134. Epub 2015 Jul 22. PMID 26202996
- [Background] Gross PR. Is pain sensitivity associated with dental avoidance? Behav Res Ther. 1992 Jan;30(1):7-13. doi: 10.1016/0005-7967(92)90090-4. PMID 1540116
- [Background] Simons, J. S., & Gaher, R. M. (2005). The Distress Tolerance Scale: Development and validation of a self-report measure. Motivation and Emotion, 29(2), 83-102. http://dx.doi.org/10.1007/s11031-005-7955-3
- [Background] Marks IM, Mathews AM. Brief standard self-rating for phobic patients. Behav Res Ther. 1979;17(3):263-7. doi: 10.1016/0005-7967(79)90041-x. No abstract available. PMID 526242
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Potter CM, Jensen D, Kinner D, Tellez M, Ismail AI, Heimberg RG. Single-session computerized cognitive behavioral therapy for dental anxiety: A case series. Clinical Case Studies. 2016;15(1):3-17.
- [Derived] Tellez M, Dunne EM, Konneker E, Zhao H, Ismail AI. Online Cognitive-Behavioural Intervention to Manage Dental Anxiety: A 12-Month Randomised Clinical Trial. Community Dent Oral Epidemiol. 2025 Oct;53(5):543-555. doi: 10.1111/cdoe.13049. Epub 2025 Jun 13. PMID 40514778

RESULTS

PARTICIPANT FLOW:
Recruitment Details: To be eligible, patients had to be between 18 and 75 years of age, fluent in spoken and written English, have scheduled a dental treatment appointment, be willing and able to give informed consent, participate responsibly in the study protocol, meet criteria for high dental anxiety based on the MDAS, and endorse at least some oral-health related impairment at the administration of a semi-structured diagnostic interview. Recruitment was carried out at Temple University School of Dentistry clinics
Pre-assignment Details: Participants were randomly assigned to one of three arms after their baseline visit was completed. Please see more information about individual arms below.
Groups:
- Psychology Intervention: Intervention was administered by psychology personnel with graduate-level training and experience in CBT (e.g., psychologists, postdoctoral fellows)
- Dental Intervention: Intervention was administered by dental staff with brief but specific training in the administration of the CBT intervention (e.g., dental assistants).
- Control: These participants were assigned to a time- and attention matched control condition, which consisted of watching an hour long nature video.
Period: Overall Study
Arm/Group | Psychology Intervention | Dental Intervention | Control
Started | 162 | 167 | 170
Intervention/Visit Day | 121 | 122 | 138
Post Appointment Debriefing | 121 | 120 | 135
1-month Follow-up | 111 | 112 | 123
3-month Follow-up | 105 | 107 | 118
Completed | 105 | 107 | 118
Not Completed | 57 | 60 | 52

BASELINE CHARACTERISTICS:
Population: 499 total participants were analyzed for this study. However, 503 were enrolled. 4 participants failed to randomize and were excluded from all analysis. All demographic and outcome information reports those 499 participants, but n=503 reported elsewhere reflects the total number of participants who were initially enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Psychology Intervention | Dental Intervention | Control | Total
Number analyzed (Participants) | 162 | 167 | 170 | 499
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.7 (15.5) | 49.3 (14.3) | 48 (14.8) | 49 (14.9)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 115 | 109 | 125 | 349
  Male | 43 | 53 | 44 | 140
  Others | 1 | 3 | 1 | 5
  Unknown/Missing | 3 | 2 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 15 | 20 | 56
  Not Hispanic or Latino | 135 | 150 | 149 | 434
  Unknown or Not Reported | 6 | 2 | 1 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3 | 6
  Asian | 8 | 8 | 6 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 2
  Black or African American | 92 | 99 | 110 | 301
  White | 47 | 43 | 39 | 129
  More than one race | 7 | 10 | 5 | 22
  Unknown or Not Reported | 6 | 6 | 5 | 17
Region of Enrollment [Number; unit: Participants]
  United States | 162 | 167 | 170 | 499
Modified Dental Anxiety Scale [Mean (Standard Deviation); unit: Score on a Scale] — The MDAS is a 5-item measure assessing fear of dental procedures, including cleaning, drilling, and local anesthetic injections; for example, "If you were about to have your tooth drilled, how would you feel?" Items are rated on a 5-point Likert-type scale ranging from 1 (not anxious) to 5 (extremely anxious). The total score ranges from 5 to 25; a score of 19 or above indicates high anxiety.
  Score on a Scale | 19.4 (3.8) | 19.4 (3.9) | 19.8 (3.1) | 19.5 (3.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Modified Dental Anxiety Scale (MDAS; Humphris et al., 1995).
Description: The MDAS is a widely used 5-item measure assessing fear of dental procedures, including cleaning, drilling, and local anesthetic injections; for example, "If you were about to have your tooth drilled, how would you feel?" Items are rated on a 5-point Likert-type scale ranging from 1 (not anxious) to 5 (extremely anxious). The total score ranges from 5 to 25; a score of 19 or above indicates high anxiety based on receiver operating characteristic analyses from previous studies.
Time Frame: The MDAS will be administered at the baseline assessment and at one- and three-month follow-ups.
Population: Overall number of participants analyzed reflects baseline enrollment numbers. 1 Month and 3 Month MDAS reports a smaller n due to participant dropout throughout the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychology Intervention | Dental Intervention | Control
Number analyzed (Participants) | 162 | 167 | 170
score on a scale
  Baseline | 19.8 (3.1) | 19.4 (3.9) | 19.4 (3.8)
  1 Month: number analyzed (Participants) | 111 | 112 | 123
  1 Month | 16.7 (4.7) | 17.2 (4.6) | 18 (4.4)
  3 Month: number analyzed (Participants) | 105 | 107 | 118
  3 Month | 15.5 (4.9) | 16.1 (4.8) | 17 (4.6)

2. Primary Outcome: Change in Rating of Dental Fear From Anxiety and Related Disorders Interview Schedule for Diagnostic and Statistical Manual -5 (DSM-5) - Adult Version (ADIS-5- Brown & Barlow, 2014)
Description: The ADIS-5 is a semi-structured interview designed to establish reliable diagnoses of the DSM-5 anxiety, mood, somatoform, and substance use disorders. To minimize participant burden, this study will utilize only the dental procedure-related section of the specific phobia module of the interview. This module includes ratings of fear and avoidance of dental procedures (0 = No fear/Never avoids to 8 = Very severe fear always avoids) as well as resultant interference (0 = None to 8 = Very severe; the latter being used to operationalize one of the inclusion criteria). For the dental phobia diagnosis, a dimensional clinical severity rating (CSR), ranging from 0 = none to 8 = very severely disturbing/disabling, will be assigned, with scores of 4 or above denoting clinical significance. All interviews will be audio-recorded. The 0-8 rating of dental fear will serve as the primary measure derived from the ADIS-5.
Time Frame: The ADIS-5 will be administered at the baseline assessment and at one- and three-month follow-ups.
Population: Note: participants who did not meet a minimum threshold of fear during the first six questions of the ADIS were not prompted to continue with the rest of the ADIS interview, including the rating of their dental fear. Participants were required to report a fear score of 4 or above on a 0-8 scale for at least one of the first six questions, which asked participants to rate how much they feared a certain common dental situation (blood from a minor cut, receiving an injection, etc.)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychology Intervention | Dental Intervention | Control
Number analyzed (Participants) | 154 | 156 | 167
score on a scale
  Baseline | 5.2 (2.0) | 5.4 (2.2) | 5.4 (2.0)
  1 Month: number analyzed (Participants) | 97 | 105 | 116
  1 Month | 4.8 (2.1) | 4.7 (2.2) | 4.8 (2.3)
  3 Month: number analyzed (Participants) | 81 | 88 | 107
  3 Month | 4.6 (1.9) | 4.4 (2.3) | 4.5 (2.2)

3. Secondary Outcome: Change in Avoidance Rating From the ADIS-5
Description: The rating of avoidance included in the specific phobia module of the ADIS-5 will be considered a secondary outcome measure. For the dental phobia diagnosis, a dimensional clinical severity rating, ranging from 0 = none to 8 = very severely disturbing/disabling, will be assigned, with scores of 4 or above denoting clinical significance.
Time Frame: baseline assessment, and at one- and three-month follow-ups.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychology Intervention | Dental Intervention | Control
Number analyzed (Participants) | 154 | 156 | 167
score on a scale
  Baseline | 4.7 (2.3) | 4.7 (2.4) | 4.7 (2.4)
  1 Month: number analyzed (Participants) | 97 | 104 | 116
  1 Month | 3.9 (2.3) | 3.9 (2.5) | 3.8 (2.5)
  3 Months: number analyzed (Participants) | 81 | 88 | 107
  3 Months | 3.7 (2.5) | 3.7 (2.5) | 3.5 (2.4)

4. Secondary Outcome: Pain Intensity Numeric Rating Scale (PI-NRS).
Description: The PI-NRS is a widely utilized 11-point self-report measure that assesses physical pain intensity on a scale ranging from 0 (no pain) to 10 (worst possible pain). Anxiety increases subjective pain experience, and therefore this scale will be used to assess the intensity of dental-related pain that participants expect to experience at their dental appointment scheduled after the dental anxiety intervention (or control), the intensity of pain they actually experienced, and the intensity of pain they expect to experience at their next similar dental appointment.
Time Frame: These ratings will be administered as part of the post-appointment debriefing interview, as well as at the 1-month and 3-month follow-ups.
Population: The question, "How much pain do you expect to experience during your next similar dental procedure?" was asked to pts as part of the PI-NRS following their dental appointment, at 1-month, and at 3-months follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Psychology Intervention | Dental Intervention | Control
Number analyzed (Participants) | 162 | 167 | 170
Participants
  Post-Appointment: number analyzed (Participants) | 104 | 107 | 126
  Post-Appointment: 0 - No pain | 21 | 16 | 12
  Post-Appointment: 1 | 8 | 10 | 4
  Post-Appointment: 2 - Mild Pain | 9 | 16 | 19
  Post-Appointment: 3 | 11 | 9 | 12
  Post-Appointment: 4 - Moderate Pain | 14 | 12 | 14
  Post-Appointment: 5 | 13 | 13 | 18
  Post-Appointment: 6 - Severe Pain | 11 | 9 | 8
  Post-Appointment: 7 | 2 | 3 | 9
  Post-Appointment: 8 - Very Severe Pain | 1 | 8 | 11
  Post-Appointment: 9 | 4 | 2 | 3
  Post-Appointment: 10 - Worst Possible Pain | 10 | 9 | 16
  1-Month Follow Up: number analyzed (Participants) | 104 | 108 | 117
  1-Month Follow Up: 0 - No pain | 9 | 12 | 11
  1-Month Follow Up: 1 | 11 | 12 | 11
  1-Month Follow Up: 2 - Mild Pain | 33 | 23 | 21
  1-Month Follow Up: 3 | 7 | 4 | 10
  1-Month Follow Up: 4 - Moderate Pain | 23 | 27 | 24
  1-Month Follow Up: 5 | 9 | 9 | 12
  1-Month Follow Up: 6 - Severe Pain | 9 | 7 | 12
  1-Month Follow Up: 7 | 0 | 4 | 7
  1-Month Follow Up: 8 - Very Severe Pain | 1 | 8 | 5
  1-Month Follow Up: 9 | 0 | 0 | 0
  1-Month Follow Up: 10 - Worst Possible Pain | 2 | 2 | 4
  3-Month Follow Up: number analyzed (Participants) | 105 | 106 | 116
  3-Month Follow Up: 0 - No pain | 12 | 14 | 9
  3-Month Follow Up: 1 | 11 | 10 | 11
  3-Month Follow Up: 2 - Mild Pain | 25 | 18 | 24
  3-Month Follow Up: 3 | 14 | 10 | 10
  3-Month Follow Up: 4 - Moderate Pain | 22 | 24 | 26
  3-Month Follow Up: 5 | 7 | 11 | 19
  3-Month Follow Up: 6 - Severe Pain | 5 | 13 | 5
  3-Month Follow Up: 7 | 2 | 2 | 4
  3-Month Follow Up: 8 - Very Severe Pain | 3 | 1 | 5
  3-Month Follow Up: 9 | 0 | 0 | 1
  3-Month Follow Up: 10 - Worst Possible Pain | 4 | 3 | 2

5. Secondary Outcome: Pain Sensitivity Index (PSI; Gross, 1992a).
Description: The PSI is a 16-item self-report measure that assesses the fearful appraisal of pain and the expected physical, psychological, and social consequences of pain. Items are rated on a scale ranging from 0 (not at all) to 7 (very much) reflecting the degree to which the item applies to the respondent. Higher scores indicate higher levels of pain sensitivity. The minimum PSI score is 0, while the maximum PSI score is 112.
Time Frame: It will be administered at baseline and the 1-month and 3-month follow-ups.
Population: Differences between number of participants analyzed and pt data reported at subsequent timepoints is due to dropout. Pts completed the MDAS and ADIS at the same time they were enrolled by study staff. However, secondary measures such as the PSI were given to pts to complete independently before the intervention visit. Participants who did not attend the intervention visit were unlikely to complete these measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychology Intervention | Dental Intervention | Control
Number analyzed (Participants) | 162 | 167 | 170
score on a scale
  Baseline: number analyzed (Participants) | 136 | 143 | 146
  Baseline | 67.3 (23.2) | 68.4 (21.6) | 68.4 (24.0)
  1 Month: number analyzed (Participants) | 104 | 108 | 116
  1 Month | 58.6 (24.3) | 63.2 (23.3) | 62.8 (25.1)
  3 Months: number analyzed (Participants) | 102 | 104 | 115
  3 Months | 55.3 (26.5) | 56.9 (23.9) | 57.9 (25.5)

6. Secondary Outcome: Distress Tolerance Scale (DTS; Simons & Gaher, 2005).
Description: The DTS is a 15-item self-report measure assessing one's perceived ability to experience and tolerate negative emotional states. This scale measures four dimensions of distress tolerance: subjective appraisal of distress, ability to tolerate emotional distress, absorption of attention by negative emotions, and regulation efforts to alleviate distress. Items are rated on a scale ranging from 1 (strongly agree) to 5 (strongly disagree). Total score range from 15 to 75, with higher scores reflecting higher levels of distress tolerance.
Time Frame: The DTS will be administered at the baseline assessment and at one- and three-month follow-ups
Population: Differences between number of participants analyzed and pt data reported at subsequent timepoints is due to dropout. Pts completed the MDAS and ADIS at the same time they were enrolled by study staff. However, secondary measures such as the DTS were given to pts to complete independently before the intervention visit. Participants who did not attend the intervention visit were unlikely to complete these measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychology Intervention | Dental Intervention | Control
Number analyzed (Participants) | 162 | 167 | 170
score on a scale
  Baseline: number analyzed (Participants) | 140 | 142 | 146
  Baseline | 45.6 (12.8) | 44.9 (12.6) | 43.7 (14.0)
  1 Month: number analyzed (Participants) | 103 | 108 | 116
  1 Month | 47.6 (13.5) | 46.3 (13.8) | 46.1 (14.4)
  3 Months: number analyzed (Participants) | 105 | 106 | 116
  3 Months | 49.3 (15.0) | 47.2 (13.7) | 47 (13.7)

7. Secondary Outcome: Fear Questionnaire Blood-Injury-Injection Subscale (FQ-BII; Marks & Mathews, 1979).
Description: The FQ-BII is a 5-item subscale of the complete FQ. It assesses the degree to which an individual avoids situations involving blood-injury-injection because of fear, including in the context of dental procedures. Items are rated on a scale ranging from 0 (would not avoid it) to 8 (would always avoid it). Total scores range from 0-40 with higher scores indicating greater phobic avoidance.
Time Frame: It will be administered at the baseline assessment and at one- and three-month follow-ups.
Population: Differences between number of participants analyzed and pt data reported at subsequent timepoints is due to dropout. Pts completed the MDAS and ADIS at the same time they were enrolled by study staff. However, secondary measures such as the FQBII were given to pts to complete independently before the intervention visit. Participants who did not attend the intervention visit were unlikely to complete these measures.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychology Intervention | Dental Intervention | Control
Number analyzed (Participants) | 162 | 167 | 170
score on a scale
  Baseline: number analyzed (Participants) | 140 | 142 | 146
  Baseline | 45.6 (12.8) | 44.9 (12.6) | 43.7 (14)
  1 Month: number analyzed (Participants) | 103 | 108 | 116
  1 Month | 47.6 (13.5) | 46.3 (13.8) | 46.1 (14.4)
  3 Months: number analyzed (Participants) | 105 | 106 | 116
  3 Months | 49.3 (15.0) | 47.2 (13.7) | 47.0 (13.7)

8. Secondary Outcome: Client Satisfaction Questionnaire (CSQ-8; Larsen et al., 1979).
Description: The CSQ-8 is used in the measurement of client/patient assessment of satisfaction with services and clinical care. It consists of 8 items rated on a 1-to-4 scale. Higher scores indicate greater satisfaction with services, with a minimum score of 8 and a maximum score of 32.
Time Frame: The CSQ-8 will be administered post-intervention (within 48 hours after the participant's dental appointment), as well as at the one- and three-month follow-ups.
Population: Differences in number of participants analyzed at each time point is due to participant drop-out throughout the study. Additionally, participants in the control condition were not administered the CSQ since the questions were not relevant to the time-and attention-matched nature video they were assigned.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychology Intervention | Dental Intervention
Number analyzed (Participants) | 105 | 108
score on a scale
  Post-Intervention | 27.3 (3.7) | 27.7 (3.7)
  1-Month: number analyzed (Participants) | 94 | 105
  1-Month | 25.9 (4.2) | 26.8 (4.3)
  3-Months: number analyzed (Participants) | 101 | 102
  3-Months | 26.4 (4.8) | 27.4 (4.3)

9. Secondary Outcome: Change in Distress and Interference Rating From the ADIS-5
Description: The rating of distress and interference included in the specific phobia module of the ADIS-5 will be considered a secondary outcome measure. For the dental phobia diagnosis, a dimensional clinical severity rating, ranging from 0 = none to 8 = very severely disturbing/disabling, will be assigned, with scores of 4 or above denoting clinical significance.
Time Frame: baseline assessment, and at one- and three-month follow-ups.
Population: Note: participants who did not meet a minimum threshold of fear during the first six questions of the ADIS were not prompted to continue with the rest of the ADIS interview, including the rating of their dental fear. Participants were required to report a fear score of 4 or above on a 0-8 scale for at least one of the first six questions, which asked participants to rate how much they feared a certain common dental situation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychology Intervention | Dental Intervention | Control
Number analyzed (Participants) | 154 | 156 | 167
score on a scale
  Baseline | 4.6 (1.6) | 4.5 (1.7) | 4.3 (1.7)
  1 Month: number analyzed (Participants) | 97 | 105 | 116
  1 Month | 4.0 (1.6) | 3.9 (1.6) | 3.7 (1.6)
  3 Month: number analyzed (Participants) | 81 | 88 | 107
  3 Month | 3.9 (1.6) | 3.6 (1.8) | 3.4 (1.5)

10. Secondary Outcome: Change in Percentage of Dentally Phobic Patients From the ADIS-5
Description: Percentage of patients who meet criteria for a specific phobia of dental procedures at baseline. We will examine whether this percentage decreases as a function of the arm of the study to which patients are assigned.
Time Frame: baseline assessment, and at one- and three-month follow-ups.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Psychology Intervention | Dental Intervention | Control
Number analyzed (Participants) | 154 | 156 | 167
Participants
  Baseline | 131 | 130 | 140
  1 Month: number analyzed (Participants) | 111 | 112 | 123
  1 Month | 72 | 73 | 84
  3 Month: number analyzed (Participants) | 105 | 107 | 118
  3 Month | 61 | 57 | 72

11. Secondary Outcome: Change in Attendance at Dental Appointments
Description: We will utilize TUKSoD's automated scheduling system (axiUm, http://www.axiumdental.com/) to collect information about dental attendance.
Time Frame: 1 year post-dental anxiety intervention
Population: Pre-Intervention = the period of 12 months preceding the participant's intervention or control visit Post-Intervention = the period of 12 months following the participant's intervention or control visit
Measure: Mean (Standard Deviation); unit: Number of Appointments
Arm/Group | Psychology Intervention | Dental Intervention | Control
Number analyzed (Participants) | 162 | 167 | 170
Number of Appointments
  Appointments No Showed (Pre-Intervention) | 0.6 (1.0) | 0.6 (1.0) | 0.7 (1.1)
  Appointments Completed (Pre-Intervention) | 6.2 (5.3) | 5.7 (4.6) | 6.2 (5.0)
  Pre-Completion Rate (Pre-Intervention) | 0.8 (0.2) | 0.8 (0.2) | 0.8 (0.2)
  Appointments Cancelled (Pre-Intervention) | 1.3 (1.9) | 1.3 (1.9) | 1.2 (1.5)
  Appointments No Showed (Post-Intervention) | 0.8 (1.2) | 0.6 (1.1) | 0.9 (1.3)
  Appointments Completed (Post-Intervention) | 5.4 (5.8) | 5.2 (5.3) | 4.6 (4.6)
  Post-Completion Rate (Post-Intervention) | 0.6 (0.3) | 0.6 (0.3) | 0.6 (0.3)
  Appointments Cancelled (Post-Intervention) | 1.7 (1.9) | 1.6 (1.9) | 1.5 (1.6)

ADVERSE EVENTS:
Time Frame: From Baseline to 3-month follow up, around 12 weeks
Description: Adverse events for this study adhere to the definition provided by ClinicalTrials.gov
Arm/Group | Psychology Intervention | Dental Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/162 | 0/167 | 0/170
Serious Adverse Events (participants affected / at risk) | 0/162 | 0/167 | 0/170
Other Adverse Events (participants affected / at risk) | 0/162 | 1/167 | 0/170
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Psychology Intervention (N=162) | Dental Intervention (N=167) | Control (N=170)
Increased anxiety post-intervention (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) — At 1-month, pt reported increased anxiety due to intervention, but was willing to continue with successive follow-ups. Pt continued attending dental apt and completed all measures. Event was assessed as "mild" and reported in MMOR.

LIMITATIONS AND CAVEATS:
Only dental treatment-seeking patients who initiated contact with the TUKSoD clinics were recruited into the study (potential for sampling bias).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/55/NCT03680755/Prot_SAP_000.pdf